CLINICAL TRIAL: NCT05301257
Title: SOSteniamoci: An Internet-based Intervention to Support Informal Caregivers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bar-Ilan University, Israel (Other)
Collaborators: Istituto Auxologico Italiano (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Noa Vilchinsky, Principal Investigator, Bar-Ilan University, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01122021
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Caregiver Burden
Keywords: informal caregiver; internet-based intervention; caregiver burden; culturally adapted; eHealth
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either control or intervention group. Participants in the control group will receive the same treatment once the intervention group is finished with the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group SOSteniamoci (Experimental): Trans-diagnostic, 8 module, 8 week long internet intervention for reducing informal caregiver burden
  Interventions: Behavioral: Intervention group SOSteniamoci
- Control Group SOSteniamoci (No Intervention): Participants in the control group will be instructed to wait. Once intervention group will be finished, participants in control group will be able to access the same intervention

INTERVENTIONS:
Behavioral: Intervention group SOSteniamoci — Intervention based on cognitive behavioural therapy principles and culturally adapted to Italian population. Intervention's main purpose is to reduce caregiver burden and increase quality of life. Intervention contains psycho-educational elements as well as examples and exercises.
  Arms: Experimental Group SOSteniamoci

SUMMARY:
The purpose of this study is to evaluate efficacy of internet intervention for informal caregivers in Italy in reducing their care-giving burden.

DETAILED DESCRIPTION:
This intervention is going to take a form of an Internet-based Intervention (IBI) consisting of eight therapeutic modules. These are the themes, as listed chronologically: Introduction, Thoughts and Acceptance, Problem Solving, Stress and relaxation, Communication, Behavioural Activation, Worry and Anxiety, Maintenance. These themes were chosen after considering topics which might be the most useful for someone in a role of an informal caregiver, considering the trans-diagnostic nature of the intervention.

Effect of the intervention will be compared against a wait-list control group. Intervention is in Italian.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or over and both gender;
2. spent at least the last couple of months providing care;
3. must have internet access and the ability to use a computer or any other compatible device;
4. must be able to complete a phone interview -

Exclusion Criteria:

1) having severe physical or mental impairments, psychiatric conditions or neurological disorders; 2) the person in need of care has a life expectancy below or approximately around 6 months; 3) not able to use a computer or an electronic device; 4) not able to complete a phone interview;

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Cargiver Burden Inventory (CBI) | Pre-treatment; Week 8; 12 months post-treatment
  This measure is used to evaluate caregiver burden. CBI contains 24 questions that are distributed within 5 facets - Time Dependency, Emotional Health, Development, Physical Health and Social Relationships. Answer options are presented on a 5-item Likert scale and ranges from from 0 ('Never') to 4 ('Nearly Always'). Total score on CBI is summed up and ranges from 0 to 96, higher score indicating higher levels of burden experienced.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS-10) | Pre-treatment; Week 8; 12 months post-treatment
  Measure will be used to evaluate levels of experienced stress. It contains 10 questions on a Likert scale ranging from 0 ('Never') to 4 ('Very Often'). Higher score indicates more severe symptoms.
The Patient Health Questionnaire (PHQ-9) | Pre-treatment; Week 8; 12 months post-treatment
  Measure will be used to evaluate depressive symptoms. It contains 9 questions that must be responded to by choosing an answer from 4-item Likert scale, where number 0 indicates 'Not at all' and 3 - 'Nearly every day'. Higher score indicates more severe symptoms.
Generalized Anxiety Disorder (GAD-7) | Pre-treatment; Week 8; 12 months post-treatment
  Measure will be used to evaluate caregiver anxiety. GAD-7 contains 7 questions that must be responded to by choosing an answer from 4-item Likert scale, where number 0 indicates 'Not at all' and 3 - 'Nearly every day'. Higher score indicates more severe symptoms.
World Health Organization (WHO-5) | Pre-treatment; Week 8; 12 months post-treatment
  This questionnaire contains 5 statements regarding individual's well-being. Each of the statements must be evaluated using 6-item Likert scale with a score of 0 indicating 'At no time' while a score of 5 - 'All the time'. Higher score indicates higher well-being.
Couple Satisfaction Inventory (CSI-4) | Pre-treatment; Week 8; 12 months post-treatment
  This questionnaire contains 4 statements regarding couple satisfaction. Each of the statements must be evaluated using a 6-item Likert scale. A higher score indicates higher couple satisfaction.
The Inclusion of Illness in the Self Scale (IIS) - Caregiver version | Pre-treatment; Week 8; 12 months post-treatment
  This scale included a set of 7 pairs of concentric circles (one labeled 'Self' and one labeled 'Other's Illness') that vary in their degree of overlap from 1 (two separate circles) to 7 (almost completely overlapping circles).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No